CLINICAL TRIAL: NCT01409434
Title: Long Term Antihypertensive Exposure and Adverse Metabolic Effects: PEAR Follow-Up Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PEAR Follow-Up
Record Dates: First submitted 2011-08-01; First posted 2011-08-04 (Estimated); Results first posted 2014-10-16 (Estimated); Last update posted 2014-10-16 (Estimated); Status verified 2014-10

CONDITIONS: Drug Induced Hyperglycemia; Secondary Hyperlipidemia
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Follow-Up Arm (Other): All patients are recruited for inclusion in the Follow-Up Arm, which is the sole arm of the study. The Follow-Up Arm includes a one time study visit in which study interventions are performed. The Follow-Up Arm involves patients from the parent study who were enrolled in the follow-up study. The intervention in the Follow-Up Arm is the Oral Glucose Tolerance Test.
  Interventions: Drug: Oral Glucose Tolerance Test

INTERVENTIONS:
Drug: Oral Glucose Tolerance Test — Administration of 75 gram oral glucose load and three plasma glucose measurements (including baseline).
  Other Names: Glucose Drink 100

SUMMARY:
This is a research study of the long term effects on blood sugar and cholesterol of blood pressure lowering medications. People are invited to participate in this research study if they participated in the Pharmacogenomic Evaluation of Antihypertensive Responses (PEAR 1, NCT00246519 or PEAR 2, NCT01203852) study and are still taking a thiazide diuretic. In PEAR, the effects on blood pressure, blood sugar, and cholesterol of the high blood pressure drugs hydrochlorothiazide and atenolol over an 18 week period were evaluated. This PEAR follow-up study will determine the effects of thiazide diuretics on blood sugar and cholesterol, but in the period since the PEAR trial. The study hypothesis is that long term exposure to thiazide diuretics results in larger increases in blood sugar and cholesterol levels than short term exposure.

DETAILED DESCRIPTION:
One in three deaths in the United States is due to cardiovascular (CV) disease. One in three US adults has hypertension, a major underlying cause of CV disease. Type 2 diabetes (T2D) and dyslipidemia are major contributors of CV morbidity and mortality among hypertensive patients. Thiazide diuretics and beta blockers are first line agents in the treatment of hypertension, but these commonly prescribed antihypertensive classes can contribute to dysfunction of glucose and lipid metabolism. In randomized controlled trials, reductions in CV outcomes due to blood pressure reduction with thiazide diuretic and beta blocker treatment are accompanied by increases in T2D incidence and exacerbation of dyslipidemia. CV morbidity and mortality resulting from persistent antihypertensive-related T2D or dyslipidemia may eventually outweigh benefits from blood pressure reduction, encouraging use of alternate antihypertensive classes especially in high risk patients. An accumulating body of published literature supports that adverse metabolic effects are induced by thiazide diuretics and beta blockers. However, the vast majority of evidence for adverse metabolic effects of antihypertensive drugs utilizes secondary analyses of data from randomized blood pressure reduction trials. To date, no published study has compared short and long term adverse metabolic effects of antihypertensive therapy in the same patient population. The Pharmacogenomic Evaluation of Antihypertensive Responses (PEAR) study is a randomized, parallel assignment trial to determine genetic influences on blood pressure response to the thiazide diuretic hydrochlorothiazide and the beta blocker atenolol. The PEAR study duration (18 weeks) is not sufficient to assess long term effects (over six months) of these antihypertensive medications. The primary aim of this study is to determine the effects of long term thiazide and beta blocker therapy on glucose and lipid metabolism in the PEAR population, in which short term effects have been assessed. Secondary analyses of this follow-up study include investigating adverse metabolic effects of long term thiazide diuretic and beta blocker therapy on insulin sensitivity and the role of potassium and uric acid in the hyperglycemic effects of thiazide diuretics.

ELIGIBILITY:
Inclusion Criteria:

* previously enrolled in PEAR study
* completed last PEAR study visit greater than 6 months prior
* receive thiazide diuretic continuously since PEAR enrollment

Exclusion Criteria:

* pregnancy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rhonda M Cooper-DeHoff, PharmD, MS, Principal Investigator — University of Florida; Jason H Karnes, PharmD, Study Director — University of Florida
Locations (1):
- University of Florida College of Pharmacy, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Follow-Up Arm: All patients are recruited for inclusion in the Follow-Up Arm, which is the sole arm of the study. The Follow-Up Arm includes a one time study visit in which study interventions are performed.
  Oral Glucose Tolerance Test: Administration of 75 gram oral glucose load and three plasma glucose measurements (including baseline).
Period: Overall Study
Arm/Group | Follow-Up Arm
Started | 44
Completed | 40
Not Completed | 4
Not completed — Protocol Violation | 4

BASELINE CHARACTERISTICS:
Population: Patients previously enrolled in the PEAR 1 or 2 study
Arm/Group | Follow-Up Arm
Number analyzed (Participants) | 44
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (10)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 41
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 20
Region of Enrollment [Number; unit: participants]
  United States | 44
Fasting Glucose [Mean (Standard Deviation); unit: mg/dL] | 91 (12)

OUTCOME MEASURES:

1. Primary Outcome: Fasting Glucose (mg/dL)
Time Frame: Fasting glucose was obtained at time 0 min.
Population: A total of 44 patients were included in the study, however 4 patients were treated with anti-diabetic medications and so were excluded from the analysis. Therefore there are a total of 40 patients that were included in the analysis.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Follow-Up Arm
Number analyzed (Participants) | 40
mg/dL | 94 (13)

2. Secondary Outcome: Oral Glucose Tolerance Test (mg/dl h)
Description: Area under the curve for the OGTT was calculated for each patient using the 3 time points (0 hour, 1 hour and 2 hour). Average value for participants is provided.
Time Frame: one oral glucose tolerance test was performed with 3 time points (0 hour, 1 hour, 2 hour)
Population: Patients that underwent an OGTT
Measure: Mean (Standard Deviation); unit: mg/dL*h
Arm/Group | Follow-Up Arm
Number analyzed (Participants) | 40
mg/dL*h | 273 (74)

3. Secondary Outcome: Triglycerides (mg/dL)
Time Frame: Triglycerides was obtained at time 0 min.
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | Follow-Up Arm
Number analyzed (Participants) | 40
mg/dl | 157 (89)

4. Secondary Outcome: Low Density Lipoprotein (mg/dL)
Time Frame: Low Density Lipoprotein was obtained at time 0 min.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Follow-Up Arm
Number analyzed (Participants) | 40
mg/dL | 117 (36)

5. Secondary Outcome: High Density Lipoprotein (mg/dL)
Time Frame: High Density Lipoprotein was obtained at time 0 min.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Follow-Up Arm
Number analyzed (Participants) | 40
mg/dL | 52 (17)

ADVERSE EVENTS:
Time Frame: 3 hour study visit
Description: Subjects were monitored over the single 3 hour study visit.
Arm/Group | Follow-Up Arm
Serious Adverse Events (participants affected / at risk) | 0/44
Other Adverse Events (participants affected / at risk) | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No